CLINICAL TRIAL: NCT02530684
Title: Study of Various Insoles in Patients With Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Brigitte Jolles, MD, Professor, University of Lausanne Hospitals
Other Study IDs: 271/14
Record Dates: First submitted 2015-07-02; First posted 2015-08-21 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Foot Orthoses

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Knee osteoarthritis: Patients with knee osteoarthritis
  Interventions: Other: insole
- Control participants: Individuals without signs of knee osteoarthritis
  Interventions: Other: insole

INTERVENTIONS:
Other: insole — Insoles available on the market without prescription

SUMMARY:
It is critical to improve our understanding of knee osteoarthritis and to design better therapeutic options for this disease. The function of the knee during walking is an important factor in the development and progression of the disease. Many models of insoles that can be inserted in regular shoes with the objectives of improving the function of the knee are available on the market without prescription. Prior studies on these insoles failed to report clear benefits for the patients, mainly because the results varied strongly between persons. Walking is a complex tasks and it is well known that everybody develops his/her individual way of walking (ie., there are subtle but very important differences in the function of the knee). This observation and the fact that patient responses could vary between individuals suggest that using the same standard insoles with all patients might not be appropriated. This further suggests that care could be greatly improved if it was possible to identify patients that would respond positively to a model of insoles. Unfortunately, while several randomized controlled trials were conducted on these insoles for knee osteoarthritis, there is a paucity of data regarding their effects on the ambulatory function of the knee. Therefore, this study aims to improve the understanding regarding the effects of insoles freely available on the market in terms of knee mechanics during walking and its relation with quality of life. This study will test the hypotheses that (i) insoles have an effect on the static and dynamic lower-limb function and (ii) that benefits perceived by the patients are related to the mechanical effects produced by the insoles.

ELIGIBILITY:
PATIENTS WITH KNEE OSTEOARTHRITIS

Inclusion Criteria:

* Knee x-ray with less than a year
* Medial compartment knee osteoarthritis
* Varus knee between 0 and 10 degrees

Exclusion Criteria:

* Neurological impairments
* Prior lower-limbs surgery
* Joint injection during the last six months
* Convergent patella

CONTROL SUBJECTS

Inclusion Criteria:

* No lower-limbs or spine osteoarthritis
* No pain during ambulation

Exclusion Criteria:

* Neurological impairments
* Prior lower-limbs surgery or current treatments

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis and control subjects
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
knee function questionnaire | Week 2 following enrollment
knee function questionnaire | week 6 following enrollment
knee function questionnaire | week 8 following enrollment
knee function questionnaire | week 12 following enrollment
knee function questionnaire | week 14 following enrollment
knee function questionnaire | week 18 following enrollment

SECONDARY OUTCOMES:
quality of life questionnaire (EQ-5D) | Week 2, 6, 8, 12, 14 and 18 following enrollment
  EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Jolles, Pr, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland